CLINICAL TRIAL: NCT06062654
Title: Ultrasound-guided Hydrodistension in Patients With Adhesive Capsulitis: a Randomized Interventional Study Aimed at Evaluating the Efficacy of Hospital-assisted Rehabilitation Treatment Compared to Home-based Rehabilitation Treatment
Brief Title: Ultrasound-guided Hydrodistension in Patients With Adhesive Capsulitis
Acronym: CAVD21
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAVD21
Record Dates: First submitted 2023-08-31; First posted 2023-10-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Adhesive Capsulitis
Keywords: Shoulder; Adhesive Capsulitis; Ultrasound
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital-assisted Rehabilitation Treatment (Experimental): Patients in the experimental group will undergo 10 sessions (about 2 each week) of rehabilitation treatment at the outpatient clinics of the U.O. Physical Medicine and Rehabilitation Unit of the Rizzoli Orthopedic Institute. The rehabilitation protocol consists of a series of commuting exercises and passive/active mobilization exercises of the glenohumeral joint.
  Interventions: Other: Hospital-assisted Rehabilitation; Other: Home-based Rehabilitation
- Home-based Rehabilitation Treatment (Active Comparator): Patients in the experimental group will have 10 sessions (about 2 each week) of rehabilitation treatment with exercises to be performed self-assisted at home. The rehabilitation protocol consists of a series of commuting exercises and passive/active mobilization exercises of the glenohumeral joint
  Interventions: Other: Hospital-assisted Rehabilitation; Other: Home-based Rehabilitation

INTERVENTIONS:
Other: Hospital-assisted Rehabilitation — Patients are assisted by a physical therapist to perform commuting exercises and active and passive mobilization of the glenohumeral joint in anterior elevation, external rotation, internal rotation, retroposition and abduction.
Other: Home-based Rehabilitation — Patients were educated by a physical therapist to perform commuting exercises and active and passive mobilization of the glenohumeral joint in anterior elevation, external rotation, internal rotation, retroposition, and abduction, which they perform at home independently.

SUMMARY:
The present study aims to compare the efficacy of assisted rehabilitation treatment, in terms of improvement of pain and shoulder articulation, in patients with stage 2 adhesive capsulitis compared with unassisted home rehabilitation treatment. This evaluation is performed following the glenohumeral capsular hydrodistension procedure performed under ultrasound monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged between 18 and 65 years;
* Stage 2 adhesive capsulitis of the shoulder, with diagnosis made by clinical, radiographic evaluation in two projections (antero-posterior, lateral) and ultrasound.

Exclusion Criteria:

* Patients unable to give consent;
* Pregnant women;
* Patients with poly-drug allergies (anesthetics, corticosteroids); 3.
* Patients with other conditions with similar clinical picture (calcific tendinopathy, glenohumeral arthrosis, rotator cuff injury, etc...).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | Baseline (0 months)
  It consists of a self-administered questionnaire with values from 0 to 130 (0 non-painful and granted shoulder activity, 130 painful and non-granted shoulder activity) consisting of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions about the severity of the patient's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty the patient has with various activities of daily living that require the use of the upper extremities.
Shoulder Pain and Disability Index (SPADI) | 2 months
  It consists of a self-administered questionnaire with values from 0 to 130 (0 non-painful and granted shoulder activity, 130 painful and non-granted shoulder activity) consisting of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions about the severity of the patient's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty the patient has with various activities of daily living that require the use of the upper extremities.
Shoulder Pain and Disability Index (SPADI) | 4 months
  It consists of a self-administered questionnaire with values from 0 to 130 (0 non-painful and granted shoulder activity, 130 painful and non-granted shoulder activity) consisting of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions about the severity of the patient's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty the patient has with various activities of daily living that require the use of the upper extremities.
Shoulder Pain and Disability Index (SPADI) | 6 months
  It consists of a self-administered questionnaire with values from 0 to 130 (0 non-painful and granted shoulder activity, 130 painful and non-granted shoulder activity) consisting of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions about the severity of the patient's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty the patient has with various activities of daily living that require the use of the upper extremities.

SECONDARY OUTCOMES:
Disability of the Arm, Shoulder and Hand (DASH) | Baseline (0 months)
  It consists of a questionnaire self-completed of more than 30 questions, with values from 0 to 100 (0 shoulder activity granted, no disability, 100 shoulder activity not granted, complete disability) prepared to measure function and symptoms in patients with any musculoskeletal impairment of the upper extremity. The questions refer to the ability to perform certain actions in the last week and the symptoms that arose while performing these actions.
Disability of the Arm, Shoulder and Hand (DASH) | 2 months
  It consists of a questionnaire self-completed of more than 30 questions, with values from 0 to 100 (0 shoulder activity granted, no disability, 100 shoulder activity not granted, complete disability) prepared to measure function and symptoms in patients with any musculoskeletal impairment of the upper extremity. The questions refer to the ability to perform certain actions in the last week and the symptoms that arose while performing these actions.
Disability of the Arm, Shoulder and Hand (DASH) | 4 months
  It consists of a questionnaire self-completed of more than 30 questions, with values from 0 to 100 (0 shoulder activity granted, no disability, 100 shoulder activity not granted, complete disability) prepared to measure function and symptoms in patients with any musculoskeletal impairment of the upper extremity. The questions refer to the ability to perform certain actions in the last week and the symptoms that arose while performing these actions.
Disability of the Arm, Shoulder and Hand (DASH) | 6 months
  It consists of a questionnaire self-completed of more than 30 questions, with values from 0 to 100 (0 shoulder activity granted, no disability, 100 shoulder activity not granted, complete disability) prepared to measure function and symptoms in patients with any musculoskeletal impairment of the upper extremity. The questions refer to the ability to perform certain actions in the last week and the symptoms that arose while performing these actions.
Visual Analogue Scale (VAS) | Baseline (0 months)
  One-dimensional scale, with values from 0 to 10 (0 no pain, 10 high pain) assessing pain intensity.
Visual Analogue Scale (VAS) | 2 months
  One-dimensional scale, with values from 0 to 10 (0 no pain, 10 high pain) assessing pain intensity.
Visual Analogue Scale (VAS) | 4 months
  One-dimensional scale, with values from 0 to 10 (0 no pain, 10 high pain) assessing pain intensity.
Visual Analogue Scale (VAS) | 6 months
  One-dimensional scale, with values from 0 to 10 (0 no pain, 10 high pain) assessing pain intensity.
American Shoulder and Elbow Scale (ASES) | Baseline (0 months)
  It consists of a questionnaire, with values from 0 to 100 (0 non-painful shoulder joint, granted, 100 non-granted shoulder joint, complete disability), on limitations in activities of daily living, one part patient self-assessment and one by the specialist.
American Shoulder and Elbow Scale (ASES) | 2 months
  It consists of a questionnaire, with values from 0 to 100 (0 non-painful shoulder joint, granted, 100 non-granted shoulder joint, complete disability), on limitations in activities of daily living, one part patient self-assessment and one by the specialist.
American Shoulder and Elbow Scale (ASES) | 4 months
  It consists of a questionnaire, with values from 0 to 100 (0 non-painful shoulder joint, granted, 100 non-granted shoulder joint, complete disability), on limitations in activities of daily living, one part patient self-assessment and one by the specialist.
American Shoulder and Elbow Scale (ASES) | 6 months
  It consists of a questionnaire, with values from 0 to 100 (0 non-painful shoulder joint, granted, 100 non-granted shoulder joint, complete disability), on limitations in activities of daily living, one part patient self-assessment and one by the specialist.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Tasto JP, Elias DW. Adhesive capsulitis. Sports Med Arthrosc Rev. 2007 Dec;15(4):216-21. doi: 10.1097/JSA.0b013e3181595c22. PMID 18004221
- [Background] Hannafin JA, Chiaia TA. Adhesive capsulitis. A treatment approach. Clin Orthop Relat Res. 2000 Mar;(372):95-109. PMID 10738419
- [Background] Boyle-Walker KL, Gabard DL, Bietsch E, Masek-VanArsdale DM, Robinson BL. A profile of patients with adhesive capsulitis. J Hand Ther. 1997 Jul-Sep;10(3):222-8. doi: 10.1016/s0894-1130(97)80025-7. PMID 9268913
- [Background] Balci N, Balci MK, Tuzuner S. Shoulder adhesive capsulitis and shoulder range of motion in type II diabetes mellitus: association with diabetic complications. J Diabetes Complications. 1999 May-Jun;13(3):135-40. doi: 10.1016/s1056-8727(99)00037-9. PMID 10509873
- [Background] Wohlgethan JR. Frozen shoulder in hyperthyroidism. Arthritis Rheum. 1987 Aug;30(8):936-9. doi: 10.1002/art.1780300815. PMID 3498494
- [Background] Griesser MJ, Harris JD, Campbell JE, Jones GL. Adhesive capsulitis of the shoulder: a systematic review of the effectiveness of intra-articular corticosteroid injections. J Bone Joint Surg Am. 2011 Sep 21;93(18):1727-33. doi: 10.2106/JBJS.J.01275. No abstract available. PMID 21938377
- [Background] BLOCKEY NJ, WRIGHT JK, KELLGREN JH. Oral cortisone therapy in periarthritis of the shoulder; a controlled trial. Br Med J. 1954 Jun 26;1(4877):1455-7. doi: 10.1136/bmj.1.4877.1455. No abstract available. PMID 13160496
- [Background] De Carli A, Vadala A, Perugia D, Frate L, Iorio C, Fabbri M, Ferretti A. Shoulder adhesive capsulitis: manipulation and arthroscopic arthrolysis or intra-articular steroid injections? Int Orthop. 2012 Jan;36(1):101-6. doi: 10.1007/s00264-011-1330-7. Epub 2011 Aug 11. PMID 21833684
- [Background] Eustace JA, Brophy DP, Gibney RP, Bresnihan B, FitzGerald O. Comparison of the accuracy of steroid placement with clinical outcome in patients with shoulder symptoms. Ann Rheum Dis. 1997 Jan;56(1):59-63. doi: 10.1136/ard.56.1.59. PMID 9059143
- [Background] Tobola A, Cook C, Cassas KJ, Hawkins RJ, Wienke JR, Tolan S, Kissenberth MJ. Accuracy of glenohumeral joint injections: comparing approach and experience of provider. J Shoulder Elbow Surg. 2011 Oct;20(7):1147-54. doi: 10.1016/j.jse.2010.12.021. Epub 2011 Apr 13. PMID 21493103
- [Background] Daley EL, Bajaj S, Bisson LJ, Cole BJ. Improving injection accuracy of the elbow, knee, and shoulder: does injection site and imaging make a difference? A systematic review. Am J Sports Med. 2011 Mar;39(3):656-62. doi: 10.1177/0363546510390610. Epub 2011 Jan 21. PMID 21257847
- [Background] Patel DN, Nayyar S, Hasan S, Khatib O, Sidash S, Jazrawi LM. Comparison of ultrasound-guided versus blind glenohumeral injections: a cadaveric study. J Shoulder Elbow Surg. 2012 Dec;21(12):1664-8. doi: 10.1016/j.jse.2011.11.026. Epub 2012 Mar 23. PMID 22445159
- [Background] Bryant M, Gough A, Selfe J, Richards J, Burgess E. The effectiveness of ultrasound guided hydrodistension and physiotherapy in the treatment of frozen shoulder/adhesive capsulitis in primary care: a single centre service evaluation. Shoulder Elbow. 2017 Oct;9(4):292-298. doi: 10.1177/1758573217701063. Epub 2017 May 17. PMID 28932287
- [Background] Ladermann A, Piotton S, Abrassart S, Mazzolari A, Ibrahim M, Stirling P. Hydrodilatation with corticosteroids is the most effective conservative management for frozen shoulder. Knee Surg Sports Traumatol Arthrosc. 2021 Aug;29(8):2553-2563. doi: 10.1007/s00167-020-06390-x. Epub 2021 Jan 9. PMID 33420809
- [Background] Song A, Higgins LD, Newman J, Jain NB. Glenohumeral corticosteroid injections in adhesive capsulitis: a systematic search and review. PM R. 2014 Dec;6(12):1143-56. doi: 10.1016/j.pmrj.2014.06.015. Epub 2014 Jul 1. PMID 24998406
- [Background] Koh ES, Chung SG, Kim TU, Kim HC. Changes in biomechanical properties of glenohumeral joint capsules with adhesive capsulitis by repeated capsule-preserving hydraulic distensions with saline solution and corticosteroid. PM R. 2012 Dec;4(12):976-84. doi: 10.1016/j.pmrj.2012.06.006. Epub 2012 Aug 30. PMID 22939238
- [Background] Park KD, Nam HS, Kim TK, Kang SH, Lim MH, Park Y. Comparison of Sono-guided Capsular Distension with Fluoroscopically Capsular Distension in Adhesive Capsulitis of Shoulder. Ann Rehabil Med. 2012 Feb;36(1):88-97. doi: 10.5535/arm.2012.36.1.88. Epub 2012 Feb 29. PMID 22506240
- [Background] Oh JH, Oh CH, Choi JA, Kim SH, Kim JH, Yoon JP. Comparison of glenohumeral and subacromial steroid injection in primary frozen shoulder: a prospective, randomized short-term comparison study. J Shoulder Elbow Surg. 2011 Oct;20(7):1034-40. doi: 10.1016/j.jse.2011.04.029. Epub 2011 Aug 4. PMID 21816628
- [Background] Zappia M, Di Pietto F, Aliprandi A, Pozza S, De Petro P, Muda A, Sconfienza LM. Multi-modal imaging of adhesive capsulitis of the shoulder. Insights Imaging. 2016 Jun;7(3):365-71. doi: 10.1007/s13244-016-0491-8. Epub 2016 Apr 23. PMID 27107871
- [Background] DePalma AF. The classic. Loss of scapulohumeral motion (frozen shoulder). Ann Surg. 1952;135:193-204. Clin Orthop Relat Res. 2008 Mar;466(3):552-60. doi: 10.1007/s11999-007-0101-7. Epub 2008 Feb 10. No abstract available. PMID 18264843
- [Background] Do JG, Hwang JT, Yoon KJ, Lee YT. Correlation of Ultrasound Findings With Clinical Stages and Impairment in Adhesive Capsulitis of the Shoulder. Orthop J Sports Med. 2021 May 10;9(5):23259671211003675. doi: 10.1177/23259671211003675. eCollection 2021 May. PMID 33997079
- [Background] Tandon A, Dewan S, Bhatt S, Jain AK, Kumari R. Sonography in diagnosis of adhesive capsulitis of the shoulder: a case-control study. J Ultrasound. 2017 Aug 21;20(3):227-236. doi: 10.1007/s40477-017-0262-5. eCollection 2017 Sep. PMID 28900523
- [Background] Chan HBY, Pua PY, How CH. Physical therapy in the management of frozen shoulder. Singapore Med J. 2017 Dec;58(12):685-689. doi: 10.11622/smedj.2017107. PMID 29242941
- [Background] Page MJ, Green S, Kramer S, Johnston RV, McBain B, Chau M, Buchbinder R. Manual therapy and exercise for adhesive capsulitis (frozen shoulder). Cochrane Database Syst Rev. 2014 Aug 26;2014(8):CD011275. doi: 10.1002/14651858.CD011275. PMID 25157702
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Derived] Vita F, Gualtierotti R, Miceli M, Tedeschi R, Origlio F, Cavallo M, Galletti S, Stella SM, Guerra E, Donati D, Faldini C. Fibro-adhesive Bursitis: A Novel Sonographic Finding in Adhesive Capsulitis Patients and a Proposal of Management. Rheumatol Ther. 2024 Dec;11(6):1519-1532. doi: 10.1007/s40744-024-00716-8. Epub 2024 Sep 12. PMID 39264535